CLINICAL TRIAL: NCT01446900
Title: Rituximab-2cda and Prolongation of Therapy With Rituximab Alone in Chronic Lymphocytic Leukaemia and Small Lymphocytic Lymphoma
Brief Title: R-2cda and Prolongation of Therapy With Rituximab Alone in Chronic Lymphocytic Leukaemia and Small Lymphocytic Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low rate in patient accrual
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEO S523/110; 2010-018519-14 (EudraCT Number)
Record Dates: First submitted 2011-06-15; First posted 2011-10-05 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2017-12

CONDITIONS: Chronic Lymphocytic Leukaemia; Small Lymphocytic Lymphoma
Keywords: Rituximab; Cladribine; Chronic Lymphocytic Leukaemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Cladribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab cladribine (Experimental)
  Interventions: Drug: Rituximab; Drug: Cladribine

INTERVENTIONS:
Drug: Rituximab — 375mg/mq, IV on day 1 of each 28 day cycle for 4 cycles. 375 mg/mq IV every 2 months for a total of 8 administrations as additional infusions for patients, who achieve a partial response or complete response after the therapy with R- 2-CdA.
  Other Names: Mabthera
Drug: Cladribine — 0,1 mg/Kg, SC from day 1 to day 5 of each 28 day cycle for 4 cycles.
  Other Names: Litak

SUMMARY:
The objective of this study is to confirm the efficacy of the association of R-2cda in patients affected by Chronic Lymphocytic Leukaemia and Small Lymphocytic Lymphoma and of evaluating the efficacy of prolongation of therapy with additional infusions of Rituximab alone in increasing and prolonging the duration of the response.

DETAILED DESCRIPTION:
Chronic Lymphocytic Leukaemia (CLL) is a lymphoproliferative disorder characterized by the progressive accumulation of monoclonal peripheral B cells in bone marrow, peripheral blood and lymphoid tissues. Median survival is about 10 years. It is now clear that front line therapy for a patient with CLL requiring treatment should be the association of purine analogue and rituximab with or without cyclophosphamide. Concerning the choice of the purine analogue, similar results have been obtained by using cladribine instead of fludarabine. Although cladribine is less commonly used, the direct comparison between the two analogues for what concerns efficacy and toxicity, has confirmed the same profile of the two drugs. Encouraging results have been obtained using the monoclonal antibody in association with the purine analogue.

The utilization of rituximab as a maintenance therapy could improve the response in cases of persistence of minimal residual disease as well as delay the insurgence of relapses thus increasing the DFS.

The objective of this study is to confirm the efficacy of the association of R-2cda and of evaluating the efficacy of prolongation of therapy with additional infusions of Rituximab alone in increasing and prolonging the duration of the response. The results of this study will be compared with existing clinical results from a group of 42 pts already treated as standard with R-2cda without additional rituximab infusions.

Patients enrolled in the study will receive 4 cycles of R-2-CdA therapy. Patients, who achieve a partial response or complete response after the therapy with R- 2-CdA, will prolong therapy with Rituximab. The therapy will begin 3 months after the end of the induction therapy and patients will receive one administration every 2 months for a total of 8 administrations.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Patients affected by CLL / SLL
* Presence of active disease defined as the presence of one of the following:

Disease related symptoms (weight loss >10% in the last 6 months, fever >38° C for 2 weeks without evidence of infection, or marked asthenia, or profuse sweating without evidence of infection) Massive nodes (at least 10 cm in longest diameter) or progressive or symptomatic lymphadenopathy Massive (at least 6 cm below left costal margin) or progressive or symptomatic splenomegaly Progressive lymphocytosis (increased >50% in 2 months) or lymphocyte doubling time < 6 months Evidence of progressive bone marrow insufficiency seen as evidence of or worsening of anemia and or thrombocytopenia Autoimmune anemia and or thrombocytopenia that is poorly responsive to corticosteroids or other standard therapy

Exclusion Criteria:

* Age < 18 years
* Patients with cardiac, pulmonary, neurological, psychiatric or serious metabolic conditions not related to CLL / SLL
* Altered hepatic function (bilirubin, GOT, GPT, or gammaGT > 2 times upper limit of normal) not attributable to CLL / SLL
* Altered renal function (creatinine > 1,5 times upper limit of normal)
* Patients with serious active infections
* Pregnancy and/ or breastfeeding
* Patients with positive serology for HBSAG or HBCAB without evaluation by a hepatologist
* Patients with positive serology for HIV
* Life expectancy of less than 12 months
* Not taking any other experimental drugs
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Cladribine (2CdA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Response to treatment | at month 17
  response will be evaluated according to Hallek criteria and definitions

SECONDARY OUTCOMES:
Duration of response | Every 6 months in the first year of follow-up and every 12 months afterwards until disease progression
  Duration of response Every 6 months in the first year of follow-up and every 12 months since second year until PD

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Martinelli, MD, Study Chair — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy

REFERENCES:
- [Background] Bertazzoni P, Rabascio C, Gigli F, Calabrese L, Radice D, Calleri A, Gregato G, Negri M, Liptrott SJ, Bassi S, Nassi L, Sammassimo S, Laszlo D, Preda L, Pruneri G, Orlando L, Martinelli G. Rituximab and subcutaneous cladribine in chronic lymphocytic leukemia for newly diagnosed and relapsed patients. Leuk Lymphoma. 2010 Aug;51(8):1485-93. doi: 10.3109/10428194.2010.495799. PMID 20578816
- [Background] Del Poeta G, Del Principe MI, Buccisano F, Maurillo L, Capelli G, Luciano F, Perrotti AP, Degan M, Venditti A, de Fabritiis P, Gattei V, Amadori S. Consolidation and maintenance immunotherapy with rituximab improve clinical outcome in patients with B-cell chronic lymphocytic leukemia. Cancer. 2008 Jan 1;112(1):119-28. doi: 10.1002/cncr.23144. PMID 17999417